CLINICAL TRIAL: NCT05481840
Title: The (Cost)Effect of Continence Material With Sensor for People With Profound Intellectual and Multiple Disabilities: Client-based Continence Care by Innovation
Brief Title: The (Cost)Effect of Smart Diaper Continence Care for People With Profound Intellectual and Multiple Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Academy Het Dorp (Other)
Collaborators: Tilburg University (Other); Stichting Trimbos-Instituut (Other); Maastricht University (Other); s Heeren Loo Zorggroep (Unknown); Esdégé-Reigersdaal (Unknown); Lunet (Unknown); Siza (Unknown); Zozijn (Unknown)
Responsible Party: Principal Investigator, Brigitte Boon, Director, Academy Het Dorp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AHD19.022; 80-85300-98-19110 (Other Grant/Funding Number: ZonMw); NL72751.091.20 (Other: CCMO)
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Incontinence
Keywords: Incontinence; healthcare technology; smart diaper; profound and intellectual disabilities; leakages; quality of life; cost-effectiveness
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial with a intervention group and waiting list group.
  Six organization will participate. They will be divided into one of the three couples. Within this couple randomization will take place at organization level, resulting in one organization receiving the intervention and a parallel group continuing regular continence care. The couples will start the research consecutively, after the previous couple finished the research (hence stepped). Due to the nature of the intervention (smart continence products) the randomization is not blinded.
Who Masked: Outcomes Assessor
Masking Description: Participants, care provider and investigator are not blinded, this is impossible concerning the nature of the intervention.
  Outcome assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receiving smart continence care by the use of continence material with sensor, in which their care professionals receive a notification when change is needed.
  Interventions: Device: Continence material with sensor
- Waiting list group (No Intervention): Will continue regular continence care as received by their care professionals. After data collection is finalized, they will receive smart continence care.

INTERVENTIONS:
Device: Continence material with sensor — Healthcare organizations are prepared for the use of smart continence care (for the intervention condition) using specially developed implementation guideline. They receive training, including how to apply continence material (only provided to intervention condition).
  Each participating location will use the product for 12 weeks. Correct size and absorption level will be determined for each participant. The optimize the result, this can change. Evaluation meetings with the caregivers, supplier and researcher will be held. Resulting in suggestions for alterations in continence care provided or products used, or giving indications that a team needs support in any way to foster the implementation.
  After 12 weeks, the implementation guidance from the research group will be phased out.
  The waiting list group will continue their continence care as usual during data collection period. Thereafter they will receive support for implementing smart continence care.
  Other Names: Abena Nova with Medisens, Abena Nova, Nova
  Arms: Intervention group

SUMMARY:
Background and study aims

Most people with profound intellectual and multiple disabilities (PIMD) use diapers. When living in a long-term care facilities, most changes of diapers are scheduled. Leading to leakages, unnecessary changes and burden to people with PIMD and their caregivers.

With the use of continence material with sensor (smart diapers) caregivers give more client-based continence care. The smart diaper (product name: Abena Nova) informs the caregivers about the saturation level of the diaper and gives a notification when change is needed or a leakage might occur. This can result in less leakages compared to regular continence care. And we will research the effect on quality of life and number of pad changes and cost effectiveness. The study also investigates the effect on the care givers.

Who can participate?

People with profound intellectual and multiple disabilities, of 18 years and older, who use diapers and live in one of the participating disability care organizations.

What does the study involve?

To investigate the effect, the disability care organization will be assigned to one of the two groups. In one group we will research the use of the smart diaper, the other group will continue their regular continence care.

Data collection started September 2021 and will continue roughly till February 2023. Research period for each location is 12 weeks, with 3 points for data collection. For the first two organization who are using the smart diaper, there is also data collection after 9 months.

Caregivers will fill out questionnaires about the quality of life, received healthcare of the participant, and keep a one week diary about the diaper changes and leakages.

To use the smart diaper, caregivers will receive training, there are meetings to optimize usage and the disability care organization will receive help from the researchers.

Possible benefits and risk of participating?

The potential benefit of participating lays within the organization itself, optimizing continence care and investigating whether this is cost effective. Any negative effect is the cost of the product and the additional time and effort it takes to start using smart diapers. For the patients the benefit is getting more optimized continence care. Any potential discomfort or risk (such as removing of swallowing the sensor) will be evaluated before the start. Any negative advice will result in not implementing the smart diaper for this person showing risk behavior. However, any of these adverse events cannot be complete diminished.

Where does the study run from?

Study is run by Academy Het Dorp, one of the researcher is also affiliated with Tranzo, Tilburg University

Who is funding the study?

ZonMW is funding the research activities. Disability care organization are themselves paying for the smart diapers.

Who is the main contact?

Vivette van Cooten, MSc Vivette.van.cooten@academyhetdorp.nl

ELIGIBILITY:
Inclusion:

* Age: ≥18 years
* Gender: male of female
* People with PIMD
* Living in a long-term care facility
* Using continence pads
* Not able to indicate the need for change of continence pads
* Caregivers see added value for use of smart continence pads

Exclusion:

* No informed consent of legal representative
* Risk of harmful behavior such as pica disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in baseline of number of leakages of continence pads per week at 12 weeks | Baseline (week 0) and at 12 weeks
  Measured by using a week long continence diary

SECONDARY OUTCOMES:
Change in number of changes of continence pads per week | Baseline (week 0), week 6, week 12 and 9 months
  Measured using a week long continence diary
Health status measured by EuroQoL (Quality of Life)-5 Dimensions (EQ-5D-5L proxy 1) of people with PIMD | Baseline (week 0), week 12 and 9 months
  Proxy (healthcare provider and if available relative) of person with PIMD fills out EuroQoL (EQ-5D-5L proxy 1) questionnaire resulting in a health status and VAS score of health of the person with PIMD.
Subjective wellbeing scores assessed by MIPQ of people with PIMD | Baseline (week 0), and week 12
  Proxy (healthcare provider and if available relative) of person with PIMD fills out Mood Interest and Pleasure questionnaire about person with PIMD, resulting in an overall score of subjective wellbeing between 0 (lowest subjective wellbeing score) and 100 (highest subjective wellbeing score).
Objective quality of life scores assessed by QOL-PMD of people with PIMD | Baseline (week 0), and week 12
  Proxy (healthcare provider and if available relative) of person with PIMD fills out Quality of Life of people with Profound Multiple Disabilities questionnaire about person with PIMD, resulting in an overall score of objective wellbeing between 0% (lowest objective quality of life score) and 100% (highest objective quality of life score).
Cost effectiveness of providing smart continence care | at week 6, week 12 and 9 months
  The cost effectiveness is measured by calculating the costs of the intervention and compare it with the financial benefits (cost reductions) due to the intervention. This includes direct healthcare costs (healthcare resource use) and related costs as laundry costs.
Cost utility of providing smart continence care | at week 12 and 9 months
  It calculates the financial costs (resulting from cost effectiveness analysis) to the additional QALY's (quality adjusted life years) gained when using smart continence care, compared to not using smart continence care. QALY is the outcome of the EUROQOL, health state. The Dutch tariff will be used to calculate the QALY from these health states.
Effect on work engagement for caregivers when using smart continence care | Baseline (week 0) and week 12
  This questionnaire includes questions about work pressure and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Boon, Prof. Dr., Principal Investigator — Academy Het Dorp, Arnhem, The Netherlands
Locations (5):
- Netherlands (5):
  - 's Heeren Loo, Amersfoort
  - Siza, Arnhem
  - Lunet, Eindhoven
  - Esdégé-Reigersdaal, Heerhugowaard
  - Zozijn, Wilp

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Cooten VJ, van Mastrigt GA, Gabrio A, Evers SM, Gielissen MF, Boon B. Smart Continence Care for People With Profound Intellectual and Multiple Disabilities Within Dutch Residential Care Facilities: Economic Evaluation Alongside a Cluster Randomized Trial. J Med Internet Res. 2025 Oct 10;27:e72017. doi: 10.2196/72017. PMID 41071602
- [Derived] van Cooten VJ, Gielissen MF, den Hollander W, van Mastrigt GA, Smeets O, Bongers IM, Boon B. Effectiveness of Smart Continence Care for People With Profound Intellectual and Multiple Disabilities: Cluster Randomized Trial. J Med Internet Res. 2025 Jul 31;27:e66389. doi: 10.2196/66389. PMID 40743514
- [Derived] van Cooten VJC, Gielissen MFM, van Mastrigt GAPG, den Hollander W, Evers SMAA, Smeets O, Smit F, Boon B. Smart Continence Care for People With Profound Intellectual and Multiple Disabilities: Protocol for a Cluster Randomized Trial and Trial-Based Economic Evaluation. JMIR Res Protoc. 2022 Nov 22;11(11):e42555. doi: 10.2196/42555. PMID 36413389